CLINICAL TRIAL: NCT01796808
Title: Autologous Fat Grafting for Pedal Fat Pad Atrophy
Brief Title: Fat Grafting for Pedal Fat Pad Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jeffrey A. Gusenoff, MD, Associate Professor of Plastic Surgery, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO12100139
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2017-04

CONDITIONS: Pedal Fat Pad Atrophy
Keywords: pedal; atrophy; fat grafting; adipose tissue
MeSH Terms: conditions — Atrophy | interventions — Anesthetics, Local; Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pathway A (Other): Screening visit followed by pedal fat grafting procedure with local anesthetic and visits at:
  1. 1 week
  2. Post op study visit 2 (1 month)
  3. Post op study visit 3 (2 month)
  4. Post op study visit 4 (6 month)
  5. Post op study visit 5 (12 month)
  6. Crossover to standard podiatry visits
  7. Study visit 6 (18 months)
  8. Study visit 7 (24 months)
  Interventions: Procedure: Pedal Fat Grafting; Other: Local anesthetic
- Pathway B (Other): Screening visit followed by:
  1. Study visit 1 (6months)
  2. Study Visit 2 (12 months)
  3. Crossover to Pathway A
  pedal fat grafting procedure and local anesthetic and visits at:
  1. 1 week
  2. Post op study visit 2 (1 month post procedure)
  3. Post op study visit 3 (2 month post procedure)
  4. Post op study visit 4 (6 month post procedure)
  5. Post op study visit 5 (12 month post procedure)
  Interventions: Procedure: Pedal Fat Grafting; Other: Local anesthetic

INTERVENTIONS:
Procedure: Pedal Fat Grafting — Fat grafting is a minimally invasive clinical procedure that has been widely used by plastic surgeons within reconstructive surgery for many years and is considered a standard of care procedure in plastic surgery. Fat tissue to be used for grafting is harvested (usually from abdomen or thighs) with a small liposuction cannula. The fat tissue is then sterilely centrifuged and allowed to decant before separating the fluid and oil layers from the fat tissue fraction. The aspirated fat is then loaded into 1cc syringes and injected into the plantar fat pad using specialized injection cannulas.
  Postoperatively, the foot will be bandaged for twenty-four hours and the subject will be advised to limit ambulation. Over the next three weeks, the patient will be instructed to wear a cushioned, supportive sneaker and participate in only activities of normal daily living, with no excessive aerobic activity.
Other: Local anesthetic — To numb the foot for the fat grafting procedure, lidocaine with epinephrine will be used. This will be injected near the posterior tibial nerve to numb the bottom of the foot.
  Local anesthetic of lidocaine with epinephrine will also be used to numb the fat graft harvest site (i.e. abdomen or thigh). This will allow a small incision to make so that tumescent solution can be injected into the area of fat graft harvest. Tumescent solution is a combination of injectible saline, epinephrine and lidocaine that causes numbness and vasoconstriction in the area where the fat will be harvested. This limits pain and bruising during the procedures. Only a very small amount of tumescent should be needed (i.e. <200ml). Only a few cc's of fat are needed for injection into the foot.
  Other Names: Lidocaine; Epinephrine

SUMMARY:
It is believed that the average person with an eighty year old life span will walk the distance of the world twice in their lifetime. The foot is comprised of a specialized fat pad to provide shock absorption and protection against breakdown. With all the walking humans do however, foot fat pad breakdown is inevitable. Trauma to the foot is compounded in the diabetic patients due to many reasons: loss of protective sensation secondary to neuropathy, reduced skin hydration, decreased soft tissue elasticity, elevated blood sugars and increased body weight to name a few. Increased foot pressure and decreased fat pad protection are the main contributing factors to callus formation, foot pain and ulcer formation.

Fat grafting is a cosmetic and reconstructive procedure that is used sometimes to help improve one's soft tissue thickness, shape and integrity. Autologous fat transplantation is a procedure using a patient's own fat that is taken by a small liposuction tube, from areas with a substantial amount of fat ( i.e. abdomen or thighs) and then transferred into the fat atrophied (decreased or worn out) area (in this case, the foot).

The investigators are performing this research in an effort to decrease foot pressure during activity and to increase the soft tissue thickness of the sole of the foot during one's lifetime. Ultimately this could help reduce foot pain, callus formation and even ulcer formation. The goal of this research is to see whether fat grafting will help decrease the prevalence of the aforementioned foot complications. The investigators hope that by using one's own fat tissue, he or she may have a longer duration of relief than by using other methods.

This is a randomized, cross-over designed study. Randomized means that patients will be enrolled by chance (like the flip of a coin) to one of two groups for the first part of the study. Cross-over means that, after the first part of the study or at one year, patients will move into the opposite group. One group will receive the fat grafting procedure with one year follow up (year A pathway) and the other will receive standard of care treatment from the patient's primary podiatrist during the first year (year B pathway). After the first year, patients will switch to the opposite year pathway for the next 12 months. Participation in this study will last approximately 24-26 months.

DETAILED DESCRIPTION:
The etiology of plantar fat pad atrophy may be age-related, due abnormal foot mechanics, steroid use, or collagen vascular disease. Displacement or atrophy of the fat pad can lead to osseous prominences in the forefoot that may be seen with painful skin lesions. Disease states, such as diabetes, may have loss of soft tissue integrity. Fat pad atrophy, regardless of the etiology, may result in significant pain, epidermal lesions, or metatarsalgia. In sensate patients, the pain can lead to emotional and physical pain, leading to productivity and financial losses.1

It is well documented that plantar pressure is directly correlated with plantar tissue thickness, with the loss of plantar fat being a fundamental mechanism for pressure related foot disorders.2,3 Autologous fat grafting to areas of plantar fat pad atrophy may reduce plantar pressures, and thus serve as a treatment for metatarsalgia, corn and callus prevention, and possibly ulcer prevention in diabetics. Plastic surgeons, with significant skills in fat grafting, can make a significant contribution.

Current treatment modalities for fat pad atrophy include silicone injections, fat injections, and other temporary fillers; however, no objective studies using autologous fat have been performed. Approximately 30 adults who experience pain from fat pad atrophy, will have the option to participate. Through a randomized, controlled, cross-over study, some patients will receive autologous fat grafting, while some will receive standard of care podiatric treatment, then cross-over to fat grafting treatment after a year. Through pedobarograph and ultrasound assessments, the focal pedal pressure and tissue thickness following treatment will be documented over two years.

The investigators hypothesize that fat grafting for areas of increased pedal pressure will help decrease foot pressure during gait and increase soft tissue thickness on the foot pad, ultimately reducing pain. The investigators also hope to demonstrate that by using autologous fat with evidence-based fat transfer techniques, results may be durable. This pilot study will help build new collaborative efforts between Foot and Ankle Surgery, Podiatry and Plastic Surgery, combining expertise in foot biomechanics with reconstructive fat grafting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to provide informed consent
* Patients with foot pain at the plantar surface of the foot near the head of the metacarpals
* 6 months post any surgical intervention to the foot
* Willing and able to comply with follow up examinations, including ultrasounds and pedobarographic studies

Exclusion Criteria:

* Age less than 18 years
* Inability to provide informed consent
* Feet with open ulcerations or osteomyelitis
* Diabetics: Type I and II
* Active infection anywhere in the body
* Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
* Known coagulopathy
* Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
* Pregnancy
* Subjects with a diagnosis of Schizophrenia or Bipolar Disorder (Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion).
* Tobacco use: Last use within 1 year per patient report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Demonstrate that autologous fat grafting decreases pedal pressure during gait and increase plantar tissue thickness. | 1-2 years
  Pressure will be measured on the pedobarograph in kg/cm2 or psi. Tissue thickness will be measured by ultrasound as mm. These measures will be performed before and after treatment with fat grafting to assess changes over time.

SECONDARY OUTCOMES:
Autologous fat grafting will demonstrate durability over time due to its biologic compatibility | 1-2 years
  Autologous fat grafting will demonstrate durability over time due to its biologic compatibility. Durability will be assessed via tissue thickness (ultrasound; mm), pressure (pedobarograph; psi), and pain score (validated Manchester Foot Pain Disability Index).

OTHER OUTCOMES:
With decreased pedal pressure and increased tissue thickness, pain and skin lesions will be reduced in patients with metatarsalgia | 1-2 years
  Pain will be assessed with the Manchester Foot Pain Disability Index, a validated foot pain questionnaire, and calluses will be assessed by physical exam and 2D photography.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Gusenoff, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Department of Plastic Surgery, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Bowling FL, Metcalfe SA, Wu S, Boulton AJ, Armstrong DG. Liquid silicone to mitigate plantar pedal pressure: a literature review. J Diabetes Sci Technol. 2010 Jul 1;4(4):846-52. doi: 10.1177/193229681000400412. PMID 20663447
- [Background] Abouaesha F, van Schie CH, Armstrong DG, Boulton AJ. Plantar soft-tissue thickness predicts high peak plantar pressure in the diabetic foot. J Am Podiatr Med Assoc. 2004 Jan-Feb;94(1):39-42. doi: 10.7547/87507315-94-1-39. PMID 14729989
- [Background] Abouaesha F, van Schie CH, Griffths GD, Young RJ, Boulton AJ. Plantar tissue thickness is related to peak plantar pressure in the high-risk diabetic foot. Diabetes Care. 2001 Jul;24(7):1270-4. doi: 10.2337/diacare.24.7.1270. PMID 11423514
- [Background] Espinosa N, Brodsky JW, Maceira E. Metatarsalgia. J Am Acad Orthop Surg. 2010 Aug;18(8):474-85. doi: 10.5435/00124635-201008000-00004. PMID 20675640
- [Background] Boulton AJ, Franks CI, Betts RP, Duckworth T, Ward JD. Reduction of abnormal foot pressures in diabetic neuropathy using a new polymer insole material. Diabetes Care. 1984 Jan-Feb;7(1):42-6. doi: 10.2337/diacare.7.1.42. PMID 6546713
- [Background] Young MJ, Cavanagh PR, Thomas G, Johnson MM, Murray H, Boulton AJ. The effect of callus removal on dynamic plantar foot pressures in diabetic patients. Diabet Med. 1992 Jan-Feb;9(1):55-7. doi: 10.1111/j.1464-5491.1992.tb01714.x. PMID 1551311
- [Background] Chairman EL. Restoration of the plantar fat pad with autolipotransplantation. J Foot Ankle Surg. 1994 Jul-Aug;33(4):373-9. PMID 7951190
- [Background] van Schie CH, Whalley A, Armstrong DG, Vileikyte L, Boulton AJ. The effect of silicone injections in the diabetic foot on peak plantar pressure and plantar tissue thickness: a 2-year follow-up. Arch Phys Med Rehabil. 2002 Jul;83(7):919-23. doi: 10.1053/apmr.2002.33058. PMID 12098150
- [Background] Pu LLQ, Coleman SR, Cui X, Ferguson REH Jr, Vasconez HC. Autologous fat grafts harvested and refined by the Coleman technique: a comparative study. Plast Reconstr Surg. 2008 Sep;122(3):932-937. doi: 10.1097/PRS.0b013e3181811ff0. PMID 18766062
- [Background] Kwan RL, Zheng YP, Cheing GL. The effect of aging on the biomechanical properties of plantar soft tissues. Clin Biomech (Bristol). 2010 Jul;25(6):601-5. doi: 10.1016/j.clinbiomech.2010.04.003. Epub 2010 May 8. PMID 20457479
- [Background] Veves A, Boulton AJ. The optical pedobarograph. Clin Podiatr Med Surg. 1993 Jul;10(3):463-70. PMID 8364849
- [Background] Walter Stephen Snyder 1909-1977. Health Phys. 1978 Jan;34(1):1-2. No abstract available. PMID 340428
- [Background] Pow DV, Morris JF. Tunicamycin, puromycin and brefeldin A influence the subcellular distribution of neuropeptides in hypothalamic magnocellular neurones of rat. Cell Tissue Res. 1992 Sep;269(3):547-60. doi: 10.1007/BF00353909. PMID 1423514
- [Background] Balkin SW. Injectable silicone and the foot: a 41-year clinical and histologic history. Dermatol Surg. 2005 Nov;31(11 Pt 2):1555-9; discussion 1560. doi: 10.2310/6350.2005.31241. PMID 16416638
- [Background] van Schie CH, Whalley A, Vileikyte L, Wignall T, Hollis S, Boulton AJ. Efficacy of injected liquid silicone in the diabetic foot to reduce risk factors for ulceration: a randomized double-blind placebo-controlled trial. Diabetes Care. 2000 May;23(5):634-8. doi: 10.2337/diacare.23.5.634. PMID 10834422
- [Background] Niermeijer P, Gips CH. Viral antibodies and the infectivity of serum in hepatitis B. N Engl J Med. 1978 Oct 26;299(17):958. doi: 10.1056/NEJM197810262991721. No abstract available. PMID 692609
- [Derived] Minteer DM, Gusenoff BR, Gusenoff JA. Fat Grafting for Pedal Fat Pad Atrophy in a 2-Year, Prospective, Randomized, Crossover, Single-Center Clinical Trial. Plast Reconstr Surg. 2018 Dec;142(6):862e-871e. doi: 10.1097/PRS.0000000000005006. PMID 30204683